CLINICAL TRIAL: NCT05289167
Title: A Phase I-II Study of High-Dose Post-Transplant Cyclophosphamide, Bortezomib and Abatacept for the Prevention of Graft-versus-Host-Disease (GvHD) Following Allogenic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Post-Transplant Cyclophosphamide, Bortezomib and Abatacept for the Prevention of Graft-versus-Host-Disease (GvHD)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-00797
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Graft-versus-host Disease
Keywords: GvHD, post transplant cyclophosphamide, abatacept
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Abatacept; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with hematological malignancies (Experimental): Participants undergoing Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) will receive a combination of cyclophosphamide, known commercially as Cytoxan®, abatacept, known as Orecia® and bortezomib commercially known as Velcade®, to reduce the rate of graft-versus-host disease (GvHD). These medications will be given for GvHD prevention during the transplant process.
  Interventions: Drug: Cyclophosphamide; Drug: Abatacept; Drug: Bortezomib

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg/kg IV over 1 hour on Day +3 and +4
  Other Names: Cytoxan®
Drug: Abatacept — Dose level 0: 10 mg/kg IV over 30 minutes on day +5
  Dose level 1: 10mg/kg IV over 30 minutes on day +5 and +14
  Dose level 2: 10mg/kg IV over 30 minutes on day +5, +14, and +28
  Other Names: Orecia®
Drug: Bortezomib — 1.3 mg/m2 IV 6 hours after graft infusion completion and 72 hours thereafter.
  Other Names: Velcade®

SUMMARY:
This is a phase I-II clinical trial. Adult subjects with hematological malignancies undergoing allogeneic HSCT from an HLA matched sibling or ≥7 out of 8 allele level HLA matched unrelated donor are eligible for the study if they meet the criteria defined in our standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Subjects will receive a standard of care conditioning regimen. Subjects will receive investigational PTCy, investigational bortezomib and investigational abatacept as GvHD prophylaxis.

DETAILED DESCRIPTION:
The study will have a phase I and phase II potions. The phase I portion will employ a 3+3 dose escalation design to define the maximum tolerated dose (MTD) of abatacept added to PTCy and bortezomib following HSCT. The phase II portion will consist of two single arm, open label, optimal 2-stage Simon design studies conducted in two separate strata for HLA matched and HLA mismatched donor transplants. Adult patients with hematological malignancies undergoing allogeneic HSCT from an HLA matched sibling or ≥7 out of 8 allele level HLA matched unrelated donor are eligible for the study if they meet the standard criteria defined in our institutional standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Subjects will receive a standard of care conditioning regimen followed by peripheral blood hematopoietic stem cells. Subjects with unrelated donors will also receive rabbit anti-thymocyte globulin (rATG). Subjects will receive investigational PTCy, investigational bortezomib and investigational abatacept as GvHD prophylaxis. The phase II portion dose of abatacept will be the MTD as determined in the phase I portion of the study. In the phase II portions, subjects will be stratified based on whether they receive a matched sibling or matched unrelated (matched) donor transplant and ≥7 out of 8, allele level matched (mismatched) unrelated donor transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Karnofsky score ≥70%
* No evidence of progressive bacterial, viral, or fungal infection
* Creatinine clearance >50 mL/min/1.72m2
* ALT and AST <3 x the upper limit of normal
* Total bilirubin <2 x the upper limit of normal (except for Gilbert's syndrome)
* Alkaline phosphatase ≤250 IU/L
* Left Ventricular Ejection Fraction (LVEF) >45%
* Adjusted Carbon Monoxide Diffusing Capacity (DLCO) >50%
* Negative HIV serology
* Negative pregnancy test: Confirmation per negative serum β-human chorionic gonadotropin (β-hCG)
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Pregnant or nursing females or women of reproductive capability who are unwilling to completely abstain from heterosexual sex or practice 2 effective methods of contraception from start of conditioning through 90 days after the last dose of study drug. A woman of reproductive capability is one who has not undergone a hysterectomy (removal of the womb), has not had both ovaries removed, or has not been post-menopausal (stopped menstrual periods) for more than 24 months in a row.
* Male subjects who refuse to practice effective barrier contraception from the start of conditioning through a minimum of 90 days after the last dose of study drug, or completely abstain from heterosexual intercourse. This must be done even if they are surgically sterilized (i.e., post-vasectomy).
* Inability to provide informed consent.
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix D), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Known allergies to any of the components of the investigational treatment regimen.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma, an in-situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Prisoners
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-03-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase I:Incidence Dose limiting toxicity (DLT) | Day+1 to Day +120
  Defined as grade 4 non-hematologic toxicity affecting the oral cavity, gastrointestinal tract, lung, heart, liver, kidney, bladder, or central nervous system.
Phase II: Grades II-IV Acute GvHD | Day+1 to Day +120
  The first day of grades II-IV acute GvHD will be recorded for that grade. This end point will be evaluated through day +120 post-transplant.

SECONDARY OUTCOMES:
Chronic GvHD | Day +1 to Day +365
  The diagnosis of chronic GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.The analysis will be based on the maximum grade of chronic GvHD
Primary graft failure | Day +1 to Day +30
  Incidence of graft failure will be calculated from date of transplant to failure for all subjects who receive a transplant and any prophylactic treatment and from date of completion of prophylactic treatment for all participants that completed treatment
Poor graft function | Day +1 to Day +30
  Incidence of poor graft function will be calculated, from date of transplant to failure for all subjects who receive a transplant and any prophylactic treatment and from date of completion of prophylactic treatment for all participants that completed treatment
Secondary graft failure | Day +1
  Evaluated after engraftment is achieved will be calculated from date of engraftment for all subjects with engraftment
Treatment-related mortality (TRM) | Day +1 to Day +730
  Analyzed based on participants that who received a transplant with any prophylactic treatment and for all subjects who received a transplant and completed prophylactic treatment.
Relapse rate (RR) | Day +1 to Day +730
  Evaluated to day +730 and will be analyzed for all subjects who received a transplant and for all transplanted subjects that completed treatment
GvHD and relapse-free survival (GRFS) | Day +1 to Day +730
  Evaluated to day +730 and considers as successes participants that are without reported GvHD III-IV acute GvHD, chronic GvHD requiring systemic therapy and have not experienced relapse or death after transplant
Overall survival (OS) | Day +1 to Day +730
  Evaluated to day +730 and considers all participants who received a transplant and for all transplanted subjects who completed prophylactic treatment

CONTACTS AND LOCATIONS:
Overall Officials: A. Samer Al-Homsi, MD, MBA, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No
Information only to approved study team